CLINICAL TRIAL: NCT06576284
Title: A 36-month Analysis of the Clinical Performance of Individualized CAD/CAM-produced Dental Implants: a Cohort Study
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Giuseppe Alexandre Romito, Vice Dean, University of Sao Paulo
Other Study IDs: 6.987.078
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Tooth Loss; Dental Implant
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Personalized implant: This is an observational, prospective, single-cohort study conducted at the University of São Paulo, São Paulo, Brazil, involving individuals who received a personalized dental implant using the iDENTICAL Dental Implant System. The aim is to evaluate the safety, efficacy, and clinical viability of these customized implants over a 36-month follow-up period.

SUMMARY:
The goal of this prospective cohort study is to evaluate the clinical performance of a new generation of customized CAD/CAM pre-fabricated root-analog dental implants over a 36-month period. The main questions it aims to answer are:

1. Are these novel implants safe, effective, and clinically viable for 36 months?
2. Do these drilling-free implants result in better post-operative outcomes compared to traditional implant techniques? Twelve patients receiving these customized implants immediately after tooth extraction will undergo clinical and radiographic examinations at 12, 24, and 36 months after prosthesis installation. The study will assess peri-implant tissue health, post-operative comfort, bone preservation, tissue integration, and implant survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Received a personalized dental implant using the iDENTICAL Dental Implant System during the previous interventional phase;
* Completed the 12-month follow-up period after implant placement in the previous interventional phase;
* Available for follow-up evaluations during the 36 months of the observational study.

Exclusion Criteria:

* Occurrence of serious complications (implant loss, infection, etc.) during the previous interventional phase;
* Development of uncontrolled medical conditions during the follow-up period;
* Inability to attend scheduled follow-up visits;
* Refusal to participate in the observational study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who received a personalized dental implant using the iDENTICAL Dental Implant System
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Radiographic success | 12 months, 24 months and 36 months
  Radiographic success, defined as the absence of peri-implant radiolucency and lack of progressive loss (> 1.7 mm) of marginal bone level (MBL) over the 36 months following implant restoration.

SECONDARY OUTCOMES:
Linear horizontal changes of peri-implant soft tissues | 12 months, 24 months and 36 months
  measured from intraoral scans at 1mm, 3mm, and 5mm below the reference gingival margin level at the time of crown placement, at 12, 24, and 36 months.
Prosthetic Level outomes | 12 months, 24 months and 36 months
  Chipping/fracture of material; Loss of retention of restoration (cementation cement fracture); Connector (Abutment) fracture; Loss/failure of restoration substrate requiring new restoration; The restoration functions as intended/satisfactorily for the subject
Peri-implant clinical parameters | 12 months, 24 months and 36 months
  Mobility (MOB)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe A Romito, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Dentistry - University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No